CLINICAL TRIAL: NCT06493617
Title: Does Cervical Mobilization Have an Effect on Hand Function in Patients With Double Crush Syndrome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Lecturer of Physical Therapy for Neurology and it's Surgery, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003943
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Double Crush Syndrome
Keywords: cervical mobilization; hand function; double crush syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): received a standard physical therapy program of nerve glide, hand strengthening exercise and mobilization
  Interventions: Other: Traditional physical therapy treatment
- Study Group (Experimental): received a cervical mobilization in addition to the standard physical therapy program for 12 sessions
  Interventions: Other: Cervical Mobilization; Other: Traditional physical therapy treatment

INTERVENTIONS:
Other: Cervical Mobilization — The technique is used to mobilize a specific cervical or upper thoracic segment (C2-C3 through T3-T4) in a posterior to anterior direction. The therapist gently applies pressure in an anteroposterior direction in the plane of the facet joint to assess mobility, resistance, end feel, and pain provocation. Gentle oscillations can be used to either inhibit pain (grades I and II) or restore motion (grades III and IV). Slight variations in depth and direction of force can be used to optimize the therapeutic effects of this technique.
  Arms: Study Group
Other: Traditional physical therapy treatment — tendon gliding exercises, median nerve gliding exercise, strengthening exercises for 60 minutes

SUMMARY:
All Double Crush Syndrome patients were assessed via VAS, BCTQ & Nerve conduction study before and after the treatment program.

DETAILED DESCRIPTION:
The patients were classified randomly into two groups, the control group received a standard physical therapy program of nerve glide, hand strengthening exercise and mobilization and the study group they received a cervical mobilization in addition to the standard physical therapy program for 12 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Thirty female patients diagnosed as Double Crush Syndrome based on the clinical diagnostic criteria of the American Academy of Neurology, (American Academy of Neurology 2019).
* Patient ages ranged from 25 to 35 years old. Patient who reported pain, hyperesthesia, and/or paresthesia at the course of median nerve distribution and upper limb.
* A Nerve Conduction Study (NCS) evidence of peripheral entrapment of median nerve at level of carpal bone "Carpal tunnel Syndrome" with a fractionated sensory nerve conduction velocity for the median nerve across the wrist of 40 m/s or less and with sensory peak latency > 3.6 ms and recordable and with motor distal latency >4.4 ms and less than 6.5ms.

Exclusion Criteria:

* Patients had Systemic disease causes double Crush Syndrome as rheumatoid arthritis (RA), thyroid disease, Diabetes mellitus (DM), Pregnant women, Patients with concomitant neurological disease as peripheral neuropathy, Patients with history of wrist surgery, fracture, or carpal tunnel injection in the last two weeks before the study, Patients who have wasting of the thenar muscles, Patients with previous surgery for CTS.
* Patients with complete conduction block on EDX or previous regular exposure to hand-held vibrating tools, Patients with Nerve Conduction Study with motor distal latency > 6.5 ms.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 4 weeks
  Used to assess degree of pain
Boston carpal tunnel syndrome questionnaire | 4 weeks
  Used to assess patients' functional ability and symptoms severity
Nerve conduction study | 4 weeks
  Used to assess sensory and motor fibers of median nerve to determine the improvement in nerve capacity and hand function

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No